CLINICAL TRIAL: NCT03178318
Title: An Observational Study Assessing the Position of Cricothyroid Membrane in Relation to Movement of Neck From Neutral to Extended Position
Brief Title: Study Assessing the Position of Cricothyroid Membrane in Relation to Movement of Neck From Neutral to Extended Position
Acronym: ULOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northampton General Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Dr C Frerk, Consultant Anaesthetist, Northampton General Hospital NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 226475
Record Dates: First submitted 2017-06-01; First posted 2017-06-06 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Difficult Intubation
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cricothyroid membrane (Other): ultrasound of the neck will identify the position of the upper and lower border of the cricothyroid membrane in extended position.
  Interventions: Procedure: ultrasound

INTERVENTIONS:
Procedure: ultrasound — ultrasound of the neck to identify the position of upper and lower border of the cricothyroid membrane.

SUMMARY:
Ability to provide oxygen to patients undergoing general anaesthesia is crucial. This is traditionally provided using face mask, supraglottic airway (breathing tube above voice box) or endotracheal tube (breathing tube in wind pipe). However in some patients it may be impossible to provide oxygen through any of these above means which can be life threatening and lead to permanent brain damage/death. One of the ideal ways of managing this emergency situation is to pass a breathing tube through a membrane in the front of the neck called cricothyroid membrane with the neck in extension position where permitted. Many studies have recommended identifying the cricothyroid membrane before general anaesthesia in high risk patients but with their head in neutral position. This study will be a pilot study to check if the cricothyroid membrane remains in the same place in neutral and extended positions.

DETAILED DESCRIPTION:
This is a non-randomised observational pilot study. The results of the study will be used to determine the size of the sample required for a planned randomised controlled trial in the future. All the volunteers will be asked to lie on a trolley with the head in neutral position- Defined as alignment of external auditory meatus (outer ear canal) to the sternal angle (prominent portion of breast bone) is horizontal. A radiologist trained in ultrasound of the neck will identify the position of upper and lower border of the cricothyroid membrane using ultrasound and then mark these borders and the centre point with a black surgical marker pen. Then the volunteer will be asked to extend the neck and the same steps will be repeated using a red surgical marker pen. The distance between the two centre points will then be measured using a calliper/ measuring scale.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18 years or above.

Exclusion Criteria:

* Age <18 years
* Inability to communicate or refuses consent
* History of problems with neck movement
* Arthritis of the neck
* Upper limb neurology

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Ultrasound measurement | 20 minutes
  The distance between the two centre points of the cricothyroid membrane when the head is kept in the neutral and extension position which is measured using the calliper or measuring device.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Frerk, Principal Investigator — Professor of Difficult Airways Society & Consultant Anaesthetist
Locations (1):
- Northampton General Hospital NHS Trust, Northampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Result] American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Practice guidelines for management of the difficult airway: an updated report by the American Society of Anesthesiologists Task Force on Management of the Difficult Airway. Anesthesiology. 2003 May;98(5):1269-77. doi: 10.1097/00000542-200305000-00032. No abstract available. PMID 12717151
- [Result] Campbell M, Shanahan H, Ash S, Royds J, Husarova V, McCaul C. The accuracy of locating the cricothyroid membrane by palpation - an intergender study. BMC Anesthesiol. 2014 Nov 22;14:108. doi: 10.1186/1471-2253-14-108. eCollection 2014. PMID 25844061
- [Result] Lamb A, Zhang J, Hung O, Flemming B, Mullen T, Bissell MB, Arseneau I. Accuracy of identifying the cricothyroid membrane by anesthesia trainees and staff in a Canadian institution. Can J Anaesth. 2015 May;62(5):495-503. doi: 10.1007/s12630-015-0326-y. Epub 2015 Jan 31. PMID 25637060
- [Result] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Result] Hochman II, Zeitels SM, Heaton JT. Analysis of the forces and position required for direct laryngoscopic exposure of the anterior vocal folds. Ann Otol Rhinol Laryngol. 1999 Aug;108(8):715-24. doi: 10.1177/000348949910800801. PMID 10453776
- [Result] Kim WH, Ahn HJ, Lee CJ, Shin BS, Ko JS, Choi SJ, Ryu SA. Neck circumference to thyromental distance ratio: a new predictor of difficult intubation in obese patients. Br J Anaesth. 2011 May;106(5):743-8. doi: 10.1093/bja/aer024. Epub 2011 Feb 24. PMID 21354999